CLINICAL TRIAL: NCT05505591
Title: Multicenter, Observational, Retrospective Cohort Study of Patients at High Risk of Bleeding Undergoing Percutaneous Coronary Intervention and Treated With Intravenous Cangrelor Infusion (ICARUS)
Brief Title: Intravenous CAngrelor in High-bleeding Risk Patients Undergoing percutaneouS Coronary Intervention (ICARUS) Registry
Acronym: ICARUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universita degli Studi di Genova (Other)
Collaborators: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Italo Porto, Full Professor of Cardiology, Universita degli Studi di Genova
Other Study IDs: ICARUS
Record Dates: First submitted 2022-08-09; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Bleeding; Coronary Artery Disease; Myocardial Infarction
Keywords: Percutaneous coronary intervention; Cangrelor; High bleeding risk; Coronary artery disease; Acute myocardial infarction
MeSH Terms: conditions — Hemorrhage; Coronary Artery Disease; Myocardial Infarction | interventions — cangrelor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- High bleeding risk: Patients treated with cangrelor who met the Academic Research Consortium (ARC) definition of high bleeding risk (HBR)
  Interventions: Drug: Cangrelor
- Non-high bleeding risk: Patients treated with cangrelor who did not meet the Academic Research Consortium (ARC) definition of high bleeding risk (HBR)
  Interventions: Drug: Cangrelor

INTERVENTIONS:
Drug: Cangrelor — Cangrelor administration during percutaneous coronary intervention for both chronic or acute coronary syndromes

SUMMARY:
The study will investigate the prevalence of high bleeding risk (HBR) features and will compare the clinical outcomes of HBR and non-HBR patients among those undergoing percutaneous coronary intervention and receiving cangrelor infusion.

DETAILED DESCRIPTION:
Cangrelor administration is currently recommended by international guidelines in patients undergoing PCI who are naïve to P2Y12 inhibitors. These recommendations are based on the large Cangrelor Versus Standard Therapy to Achieve Optimal Management of Platelet Inhibition (CHAMPION) program, which encompassed three randomized controlled trials (RCTs) enrolling both chronic and acute coronary syndromes. Consistently, the aforementioned studies showed the benefit of cangrelor in terms of ischemic events (mainly driven by a reduction of myocardial infarction - MI - and stent thrombosis - ST) in the face of an increased rate of minor bleeding. However, those RCTs were primarily focused on populations at considerable ischemic risk and with predictably low bleeding proneness, including young patients without bleeding risk features.

In the contemporary practice, however, PCI is increasingly frequent in patients at high risk of bleeding, who are not formally prevented from being administered with cangrelor by international guidelines and possibly necessitate powerful and rapid-onset platelet inhibition while undergoing complex percutaneous revascularization. The present registry was therefore conceived at the scope of collecting data on the use of cangrelor in high bleeding risk (HBR) patients undergoing contemporary PCI. Specifically, it will assess the frequency of HBR patients in a real-world cohort of individuals treated with cangrelor and will compare the clinical outcomes of HBR and non-HBR patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Cangrelor administration during percutaneous coronary intervention for both acute and chronic coronary syndromes

Exclusion Criteria:

1. Cangrelor administration as a bridge to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing percutaneous coronary intervention with cangrelor infusion will be included.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Rate of NACE | 48 hours
  A composite of cardiovascular death, myocardial infarction, stroke, definite or probable stent thrombosis and Bleeding Academic Research Consortium 2-5 bleeding

SECONDARY OUTCOMES:
Rate of MACE | 48 hours
  A composite of cardiovascular death, myocardial infarction, stroke and definite or probable stent thrombosis
Rate of cardiovascular death | 48 hours
  Cardiovascular death according to the ARC definition
Rate of myocardial infarction (periprocedural) | 48 hours
  Myocardial infarction (periprocedural) according to the 4th Universal definition
Rate of ischemic stroke | 48 hours
  An acute episode of focal or global neurological dysfunction caused by central nervous system (CNS) vascular injury as a result of infarction, involving the brain, spinal cord or retina
Rate of hemorrhagic stroke | 48 hours
  An acute episode of focal or global neurological dysfunction caused by central nervous system (CNS) vascular injury as a result of hemorrhage, involving the brain, spinal cord or retina
Rate of definite or probable stent thrombosis | 48 hours
  Definite or probable stent thrombosis according to the ARC definition
Rate of bleeding Academic Research Consortium (BARC) 2,3 and 5 bleeding | 48 hours
  Bleeding grade 2,3 and 5 according to the ARC definition
Rate of bleeding Academic Research Consortium (BARC) 3 and 5 bleeding | 48 hours
  Bleeding grade 3 and 5 according to the ARC definition
Rate of MACE | During hospital stay (up to discharge day), on average 5 days
  A composite of cardiovascular death, myocardial infarction, stroke and definite or probable stent thrombosis
Rate of cardiovascular death | During hospital stay (up to discharge day), on average 5 days
  Cardiovascular death according to the ARC definition
Rate of myocardial infarction | During hospital stay (up to discharge day), on average 5 days
  Myocardial infarction according to the 4th Universal definition
Rate of ischemic stroke | During hospital stay (up to discharge day), on average 5 days
  An acute episode of focal or global neurological dysfunction caused by central nervous system (CNS) vascular injury as a result of infarction, involving the brain, spinal cord or retina
Rate of hemorrhagic stroke | During hospital stay (up to discharge day), on average 5 days
  An acute episode of focal or global neurological dysfunction caused by central nervous system (CNS) vascular injury as a result of hemorrhage, involving the brain, spinal cord or retina
Rate of definite or probable stent thrombosis | During hospital stay (up to discharge day), on average 5 days
  Definite or probable stent thrombosis according to the ARC definition
Rate of blood transfusion | During hospital stay (up to discharge day), on average 5 days
  Blood transfusion during hospital stay

OTHER OUTCOMES:
Rate of all-cause death | 48 hours
  All-cause death
Rate of thrombolysis in myocardial infarction (TIMI) major bleeding | 48 hours
  Major bleeding according to the TIMI definition
Rate of thrombolysis in myocardial infarction (TIMI) minor bleeding | 48 hours
  Minor bleeding according to the TIMI definition
Rate of all-cause death | During hospital stay (up to discharge day), on average 5 days
  All-cause death
Rate of all-cause death | Through the longest available follow-up, an average of 1 year
  All-cause death

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Università degli Studi della Campania "Luigi Vanvitelli", Caserta
  - University of Genoa, Genova

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Benenati S, Gragnano F, Scalamera R, De Sio V, Capolongo A, Cesaro A, Annibali G, Campagnuolo S, Silverio A, Bellino M, Centore M, Schettino M, Bertero E, Caretta G, Rezzaghi M, Veneziano F, De Nardo D, De Rosa G, De Luca L, Galasso G, Menozzi A, Musumeci G, Cirillo P, Calabro P, Porto I. ICARUS score for predicting peri-procedural bleeding in patients undergoing percutaneous coronary intervention with cangrelor. Int J Cardiol. 2024 Dec 15;417:132568. doi: 10.1016/j.ijcard.2024.132568. Epub 2024 Sep 14. PMID 39284439